CLINICAL TRIAL: NCT03974672
Title: A Retrospective Study Using a T Drain Approach Treating Anastomotic Leaks After Gastrointestinal Surgery
Brief Title: A T Drain Approach Treating Anastomotic Leaks After Gastrointestinal Surgery
Acronym: TDRAIN
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, yaron rudnicki, Principal Investigator, Meir Medical Center
Other Study IDs: MMC-0340-16-CTIL
Record Dates: First submitted 2019-05-26; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Colorectal Cancer; Diverticulitis
MeSH Terms: conditions — Colorectal Neoplasms; Diverticulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T drain: Patients treated with a T drain approach
  Interventions: Procedure: Re-laparotomy
- Stoma: Patients treated with a stoma
  Interventions: Procedure: Re-laparotomy

INTERVENTIONS:
Procedure: Re-laparotomy

SUMMARY:
Assessing the use of a T drain approach for an anastomotic leak after gastrointestinal surgery. The study's aim is to retrospectively assess the safety and benefits of this approach.

DETAILED DESCRIPTION:
Assessing the use of a T drain approach for an anastomotic leak after gastrointestinal surgery. The T drain approach is inserting a latex t tube drain into the leak site of the anastomosed bowel and diverting the fecal matter. The study's aim is to retrospectively assess the safety and benefits of this approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients after elective or emergent gastrointestinal surgery with a leak in their GI anastomosis

Exclusion Criteria:

* under 18 years of age
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after elective or emergent gastrointestinal surgery with a leak in their GI anastomosis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Measuring severity of complications with the Dindo Clavien complications scale | 30 day post operation
  By using the Dindo Clavien complications scale assessment of recuperation and complications rate and severity following re-laparotomy and assessing if another surgery was avoided.

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Rudnicki, MD, Principal Investigator — Meir Medical Center Israel
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Undecided
All none identifying patients information